CLINICAL TRIAL: NCT07225166
Title: A Clinical Investigation Into the Association of an Impaired Skin Barrier and Infant and Toddler Sensitive Skin
Status: Completed | Type: Observational
Sponsor: Kenvue Brands LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CS2025SK100263
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11-07

CONDITIONS: Sensitive Skin; Non-sensitive Skin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sensitive Skin Group: * 5-8 babies that are 3 to 6 months old
  * At least 5 babies that are 7 to 12 months old
  * At least 10 toddlers that are 13 to 36 months old
  Interventions: Other: Expert Clinical Grading; Other: Instrumental Measurements; Other: Parental Questionnaires; Other: Biomarker Measurements
- Non-Sensitive Skin Group: * 5-8 babies that are 3 to 6 months old
  * At least 5 babies that are 7 to 12 months old
  * At least 10 toddlers that are 13 to 36 months old
  Interventions: Other: Expert Clinical Grading; Other: Instrumental Measurements; Other: Parental Questionnaires; Other: Biomarker Measurements

INTERVENTIONS:
Other: Expert Clinical Grading — The expert grader will separately assess each child subject's face and body (right and left volar forearms combined, right and left leg combined, torso) for each of the parameters below according to the following 4-point scales (half points are allowed):
  - Visual Dryness, Tactile Surface Roughness, Erythema.
Other: Instrumental Measurements — The following procedures will be conducted on the child subject:
  * Corneometer measurements
  * Tewameter measurements
  * Skin pH Meter measurements
Other: Parental Questionnaires — The following questionnaires will be given to the parent subject to answer:
  * Questionnaire: Reaction to Environmental, Chemical, and Mechanical Stimuli
  * Questionnaire: Medical/Family History Questionnaire
  * Questionnaire: Bathing and Skincare Routines
Other: Biomarker Measurements — The following procedures will be conducted on the child subject:
  * D-Squame skin sampling (for corneocyte visualization and lipid analysis)
  * Microbiome sampling
  * D-Squame skin sampling (for inflammatory proteins)

SUMMARY:
This is a Single center, evaluator-blinded clinical trial that intends to • Evaluate differences in TEWL measurements between parent-reported sensitive skin subjects and healthy subjects (subjects without sensitive skin) • Evaluate differences in skin capacitance between parent-reported sensitive skin subjects and healthy subjects (subjects without sensitive skin). A sufficient number of subjects pairs (comprised of a parent subject and a child subject) will be enrolled to complete the study with at least 60 subject pairs (30 subject pairs per group).

ELIGIBILITY:
Inclusion Criteria:

Subject pairs must meet all the following inclusion criteria for enrollment into the study (only one eligible child subject may be enrolled with any one parent subject).

Parent subject and child subject:

1. Generally, in good health based on medical history reported by the parent subject.
2. Intends to complete the study and is willing and able to follow the subject responsibilities and undergo necessary testing procedures (tape stripping for baby subjects) and answer multiple questionnaires.

   Child subject:
3. Males and females aged 3 months-old up to 36 months-old (inclusive), targeting to complete with:

   Sensitive Skin Cohort (cohort 1): at least 30 child subjects in the 3 months-old up to 36 months-old range with 100% HCP diagnosed sensitive skin or parent-reported sensitive skin, and as defined as parent subjects who respond "Yes" to the Yes/No question "Do you believe your child has sensitive skin?"

   Non-Sensitive Skin Cohort (cohort 2): at least 30 child subjects in the 3 months-old up to 36 months-old age range with 100% having normal skin, has never been diagnosed with sensitive skin by a HCP, and as defined as parent subjects who respond "No" to the Yes/No question "Do you believe your child has sensitive skin?"
4. Has parent-reported natural skin tone "pale/fair to light white," "white to light beige," "beige to light tan/light olive," "medium tan/medium olive to light brown," "medium brown to dark brown," "darkest brown to darkest black", with every effort made to complete with at least 1 child subject for each skin tone per cohort.

   Parent subject:
5. Is at least 18 years old.
6. Is the primary caregiver and legal guardian of the child subject and is willing and able to present proof of legal guardianship (e.g. birth certificate/hospital discharge paperwork along with valid ID of legal guardian, etc.).
7. Is able to read, write, speak, and understand English.
8. Has signed the Consent for Photo Release and ICD including a Health Insurance Portability and Accountability Act (HIPAA) disclosure.
9. Intends to complete the study and is willing and able to follow all study instructions.
10. Parent subjects must agree to discontinue child's current face/body washes and face/body lotions for 24 hours prior to their study visit.

Exclusion Criteria:

Child Subject:

1. Is using Systemic or topical over-the-counter (OTC) or prescription medications that, in the Investigator's judgement, will affect skin condition or interfere with study evaluation. (Use of acetaminophen as needed is acceptable if it was instructed by the baby's pediatrician. Child vitamins are allowed.)
2. Is using topical steroids within 2 weeks before Visit 1.
3. Has Type 1 or Type 2 diabetes(reported by the parent) or is taking insulin or another anti-diabetic medication.
4. Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including:

   1. Immunosuppressive or steroidal drugs within 2 months before Visit 1
   2. Non-steroidal anti-inflammatory drugs within 5 days before Visit 1
   3. Antihistamines within 2 weeks before Visit 1
   4. If an individual is taking one of these medication types, the individual is not considered eligible at screening. However, if a subject begins using one of these medications during the study, the Investigator should be consulted to consider the impact of the specific medication on subject safety and/or the study results.
5. Has a history of or a concurrent health/other condition/situation which may put the child subject at significant risk, confound the study results, or interfere significantly with the subject pair's participation in the study, as determined by the Investigator or designee.
6. Has a history of skin cancer.
7. Is simultaneously participating in another study involving product usage or skin sampling for the duration of the study or has participated in another study involving product usage or skin sampling within 14 days prior to Visit 1.
8. Has used new facial and body products and/or brands two weeks prior to Visit 1.
9. Is an immediate family member of the Investigator, Study Site, or Sponsor.
10. Presents with a skin condition that may confound the study results, increase risk to the subject, or influence the outcome of the study (e.g., psoriasis, eczema, atopic dermatitis, cutaneous xerosis, or active skin cancer), as determined by the Investigator or designee.

    Parent subject:
11. Is simultaneously participating in another study.
12. Is an employee/contractor of the Study Site or Sponsor or immediate family member of the PI, Study Site, or Sponsor.

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Babies aged 3 to 36 months with either having HCP-diagnosed sensitive skin or parent-reported sensitive skin.
  Babies aged 3 to 36 months who have never been diagnosed with sensitive skin by a HCP nor have parent-reported sensitive skin.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-11-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
Corneometer measurement results | Visit 1 (Day 0)
  Higher values indicate greater hydration of the skin
Tewameter measurement results | Visit 1 (Day 0)
  Lower values reflect a reduced rate of water loss (improved skin barrier function)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS North America, Inc. - Dallas Research Center, Richardson, Texas, United States

IPD SHARING:
Plan to Share IPD: No